CLINICAL TRIAL: NCT07256873
Title: Comparison of Validity and Reliability of Core Stability and Functional Capacity Assessments Using Face-to-Face and Tele-Assessment Methods in Individuals With Chronic Low Back Pain
Brief Title: Validity and Reliability of Face-to-Face and Tele-Assessment of Core Stability and Functional Capacity
Status: Recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Sherouk Labeeb, Principal Investigator, Istinye University
Other Study IDs: ISTU-PT-CLBP-2025
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Chronic Low Back Pain (CLBP)
Keywords: Chronic low back pain; Core stability; Functional capacity; Validity, Reliability; Face-to-face assessment; Tele-assessment
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic Low Back Pain: Participants diagnosed with nonspecific chronic low back pain who will undergo core stability and functional capacity assessments using two methods: (1) face-to-face clinical evaluation and (2) tele-assessment via video communication platforms.
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — This observational study compares two assessment methods used to evaluate core stability and functional capacity in individuals with chronic nonspecific low back pain. Participants undergo standardized clinical tests performed first through face-to-face assessment and then through tele-assessment using secure video communication platforms. The assessments include Plank Test, Side Plank Test, Biering-Sorensen Test, Trunk Flexor Endurance Test, Timed Up and Go (TUG), 30-Second Chair Stand Test, 1-Minute Stair Climb Test, Visual Analog Scale (VAS), and Oswestry Disability Index (ODI). No therapeutic intervention is administered; only evaluation procedures are performed.

SUMMARY:
This study aims to compare the validity and reliability of core stability and functional capacity measurements when performed face-to-face and through tele-assessment in individuals with chronic low back pain. Chronic low back pain affects a large portion of the adult population and is associated with reduced core muscle endurance, impaired postural control, and decreased functional capacity. Tele-assessment has become increasingly important, especially after the pandemic, but there is limited evidence regarding its validity and reliability for physical performance tests.

In this study, 36 individuals with nonspecific chronic low back pain will complete core stability tests (plank, side plank, Biering-Sørensen test, and trunk flexor endurance test), functional capacity tests (Timed Up and Go, 30-Second Chair Stand, and 1-Minute Stair Climb), and questionnaires including the Visual Analog Scale and the Oswestry Disability Index. Assessments will be performed by the same physiotherapist first face-to-face in the clinic, then by tele-assessment, and tele-assessment will be repeated after 5-7 days to assess test-retest reliability.

The results are expected to show whether tele-assessment provides accurate and reliable measurements compared with traditional face-to-face evaluation. The findings may support the safe and evidence-based use of tele-assessment methods in physiotherapy practice for individuals with chronic low back pain.

DETAILED DESCRIPTION:
Chronic low back pain is one of the most common musculoskeletal disorders and is associated with decreased core muscle endurance, postural control impairments, and reduced functional capacity. In clinical practice, the evaluation of core stability and functional performance is typically performed through face-to-face assessments. However, the increasing use of tele-health, particularly after the pandemic, has created the need to determine whether these assessments can be performed remotely with acceptable validity and reliability. Existing literature on tele-assessment for musculoskeletal evaluation is limited and often includes small sample sizes or insufficient test standardization.

This study will include 36 individuals with nonspecific chronic low back pain. Participants will complete a series of core stability tests (plank test, side plank test, Biering-Sørensen test, and trunk flexor endurance test), functional capacity tests (Timed Up and Go, 30-Second Chair Stand, and 1-Minute Stair Climb), and clinical scales including the Visual Analog Scale and the Oswestry Disability Index. All assessments will be administered by the same physiotherapist. The first evaluation will be conducted face-to-face in the clinic. A second evaluation will be performed through tele-assessment using a secure video-communication platform, and a third tele-assessment will be conducted 5-7 days later to measure test-retest reliability.

The study aims to compare the results obtained from face-to-face and tele-assessment methods and to determine the validity and reliability of tele-assessment for core stability and functional capacity measurements in individuals with chronic low back pain. The findings are expected to contribute to the evidence-based use of tele-assessment in physiotherapy practice and support its integration into clinical decision-making for patients who have limited access to in-person evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Must have been diagnosed with chronic (>3 months) nonspecific low back pain.
* Must be between 18 and 65 years of age.
* Must be able to independently perform activities of daily living.
* Must not have had previous surgery for low back pain.
* Must be clinically fit to safely perform the tests specified in the research protocol.
* Must have access to the necessary technology (mobile phone, tablet, or computer, internet connection) to participate in in-person and tele-assessment sessions.
* Must be willing to participate in the study and provide written consent.

Exclusion Criteria:

* History of back surgery or serious trauma.
* History of neurological, rheumatological, cardiovascular, or pulmonary disease.
* Presence of severe scoliosis, kyphosis, or other structural spinal deformities.
* Acute pain, serious musculoskeletal injury, or orthopedic problem that prevents exercise.
* Inability to perform tests safely due to vision and/or hearing loss.
* Inability to follow instructions due to psychiatric or cognitive problems.
* Lack of technological infrastructure for online interviews and tele-assessments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with nonspecific chronic low back pain who meet the inclusion criteria and are able to participate in both face-to-face and tele-assessment sessions.
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Plank Test (Forearm Plank Test) | 4 weeks
  The plank test is used to measure the endurance capacity of all trunk stabilizers, especially the abdominal muscles. It evaluates the time it takes to maintain the trunk in a neutral position for an extended period. The individual stands parallel to the floor, supported by their forearms and toes. The body should form a straight line, and the hips should not sag or rise. The maximum time the participant can maintain this position is measured with a stopwatch
Side Plank Test (Side Bridge Test) | 4 weeks
  This test is used to evaluate the endurance of the oblique abdominal muscles, quadratus lumborum, and lateral trunk stabilizers. This test focuses on lateral trunk stability. The participant lies on their side, supported by their elbows and the outer edge of their feet. The trunk should be parallel to the floor and in a straight line. The time they can maintain this position is measured. It is usually performed separately for each side and compared
Biering-Sørensen Test | 4 weeks
  This is a standard test that evaluates the isometric endurance of the lower back extensor muscles (especially the erector spinae). A relationship has been shown between trunk extensor muscle endurance and pain levels in individuals with low back pain. The participant lies prone with their hips toward the edge of a table. The pelvis is supported on the table at the level of the pelvis, and the hips and legs are fixed. The trunk is released into a horizontal position, and the duration of the individual's ability to maintain this position is measured with a stopwatch
Flexor Endurance Test (Curl-Up Test / Trunk Flexor Endurance Test) | 4 weeks
  This test is used to measure the isometric endurance of the trunk flexor muscles (especially the rectus abdominis and oblique muscles). The ability to hold the trunk in a flexed position for extended periods is assessed. The participant lies supine, knees bent 90 degrees, and hands crossed on the chest. The participant is asked to maintain a slightly raised (30°) flexed position for as long as possible. The time is measured with a stopwatch
Timed Up and Go Test | 4 weeks
  The Timed Up and Go Test test is used to assess an individual's mobility level, balance, walking speed, and functional mobility. It is also frequently used for individuals at risk of falls. The participant sits in a standard-height chair. On the command "Go," the participant: Gets up from the chair, walks 3 meters forward, returns, and sits back down. The time it takes to complete this process is measured with a stopwatch.
30-Second Chair Stand Test | 4 weeks
  This test is used to assess lower extremity muscle strength and endurance. It also provides information about the individual's level of independence in activities of daily living. The participant sits upright in a standard-height chair, arms crossed across the chest. On the command "Go," the participant is asked to get up and sit down from the chair as many times as possible within 30 seconds. A score is obtained by counting the number of times the participant stands and sits down
1-Minute Stair Climb Test | 4 weeks
  This test provides information about an individual's cardiorespiratory endurance and lower extremity muscle strength. It is particularly preferred for functional assessments based on aerobic capacity. The participant attempts to climb a standard set of stairs at their own pace for 1 minute. The number of stairs climbed at the end of the time is recorded.

SECONDARY OUTCOMES:
Visual Analog Scale | 4 weeks
  The Visual Analog Scale is a simple, valid, and reliable measurement tool used to assess individuals' subjective pain intensity. It is one of the most widely used pain assessment methods in clinical practice. The VAS is usually presented as a 10-cm-long horizontal line. The left end represents "no pain," and the right end represents "unbearable pain." The participant indicates the current pain intensity by marking a point on the line. The marked point is measured with a ruler, resulting in a score from 0 to 10
Oswestry Low Back Pain Functional Disability Index | 4 weeks
  The Oswestry Low Back Pain Functional Disability Index is an internationally recognized questionnaire used to assess the level of functional disability, particularly in individuals with low back pain. It consists of 10 sections: pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sexual life, social life, and travel. Each section is scored from 0 to 5. The total score is calculated out of 50 and converted to a percentage value.

CONTACTS AND LOCATIONS:
Locations (1):
- Kubra Kardeş, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided